CLINICAL TRIAL: NCT02612818
Title: Prevention of Adhesions During Celioscopy for Endometriosis. Impact of the Use of Anti-adhesion Treatment on Clinical Signs and Fertility at One Year
Acronym: ENDHY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ENDHY
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2017-07

CONDITIONS: Endometriosis, Adhesive
Keywords: coelioscopy
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Coelioscopy

SUMMARY:
Thus is a longitudinal, prospective, multicentric observational study performed in mainland France, among a sample of gynaecology surgeons practising at endometriosis "expert" centres.

The aim of this study is to describe, under real treatment conditions in patients suffering from endometriosis, the impact of the use of anti-adhesion treatment during celioscopy surgery on the development of clinical signs in the patients and their fertility at one year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of procreation age and who have undergone treatment for endometriosis through celioscopic surgery.
* Patients for whom spontaneous pregnancy is possible, whether or not they wish to become pregnant immediately.
* Patients accepting and able to update a questionnaire in French.
* Informed patients who agree to computerised processing of their medical data and their right of access and rectification.

Exclusion Criteria:

* Patients for whom a medical assistance programme for procreation (IVF, artificial insemination) is currently in progress.
* Patients presenting with an absolute or relative contra-indication for use of an anti-adhesion agent (severe allergic antecedents etc).
* Patients not wishing to become pregnant.
* Patients participating or having participated during the previous month in a gynaecological clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subsequent patients of procreation age having undergone a cœlioscopy for endometriosis, for whom a spontaneous pregnancy is possible, whether or not they wish to become pregnant immediately, and meeting all of the selection criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change on the clinical signs | At 2 months and one year after the baseline visit (i.e. celioscopy)
  The clinical change will be established after one year via the pain symptomatology reported by the patient, the rate of relapse (re-hospitalisation) and the rate of any eventual complications from the celioscopy (adhesions, etc.).
Fertility | One year after the baseline visit (i.e. celioscopy)
  rate of pregnancy women

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN-DEMARS, MD, Study Director — Nordic Pharma
Locations (1):
- Nordic Pharma, Paris, France